CLINICAL TRIAL: NCT03505268
Title: The Impact of Telehealthcare Intervention on Glycemic Control in Children and Adolescents With Type 1 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assuta Hospital Systems (Other)
Responsible Party: Principal Investigator, Zohar Landau, Principal Investigator, Assuta Hospital Systems
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016033
Record Dates: First submitted 2017-12-12; First posted 2018-04-23 (Actual); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Glycosylated hemoglobin A1c (HbA1c), Telemedicine
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- telemedicine intervention (Experimental): The intervention group, in addition to usual care, will get 10 telemedicine interventions by a certified nurse and dietitian who both specialize in treatment of type 1 diabetes.
  Interventions: Behavioral: Telemedicine
- usual care (No Intervention): Usual care consisted of visits to the diabetes center every three months and communication with their doctor by phone when needed.

INTERVENTIONS:
Behavioral: Telemedicine — Patients of the Intervention Group will have once biweekly telephonic intervention conversation with dietitian, specialized in diabetes and diabetes nurse. The patients of the control group will have a routine care.
  Arms: telemedicine intervention

SUMMARY:
This study evaluates the effect of telemedicine intervention program upon glycemic control in type 1 diabetes mellitus children and their parents in Israel. Half of the participants will receive the telemedicine intervention for a period of six months while the other half will receive the regular treatment then vice versa. Each group will receive in the intervention period 6 telemedicine meeting with a dietician and six telemedicine meetings with a nurse.

The investigators hypothesized that the participants that are recieving the telemedicine intervention will have a better glycemic control after 6 months.

DETAILED DESCRIPTION:
The prevalence of type 1 diabetes has been steadily increasing for the past few decades and is a relatively common chronic disease of childhood (1). Managing type 1 diabetes in young children presents unique challenges to the patient, parents, and to the pediatric health care provider. The diabetes regimen includes intensive blood glucose monitoring, multiple daily injections of insulin ,and frequent insulin dose adjustments according to the amount of carbohydrate eaten, blood sugar, and physical activity. The Diabetes Control and Complications Trail (DCCT) showed a significant link between blood glucose control and a slower onset and progression of diabetes complications, with improved glycemic control decreasing the risk of micro- and macro- vascular complication (2,3,4).

Glycosylated hemoglobin A1c (HbA1c) measures the

In the past decade a significant progress took place in therapy and treatment of diabetes. However poor glycemic control is recorded in a significant proportion of adolescents.

Telehealthcare is the use of telecommunications to deliver healthcare services and involves the remote interaction between a primary care provider and specialist. Telemedicine represents a useful and cost-effective solution to the strict follow-up required in diabetes management ,

ELIGIBILITY:
Inclusion Criteria:

diagnosed with typ1 1 diabetes for at least 6 months insulin dependent participants provided consent to participate in the study consent to use the Accu-Chek Connect diabetes management app -

Exclusion Criteria:

new onset of diabetes type 1 not specified as type 1 diabetes

-

Ages: 1 Year to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2019-05-03 (Estimated); Study Completion 2019-05-03 (Estimated)

PRIMARY OUTCOMES:
The impact of telehealthcare intervention on the change of the glycemic control in children with type 1 diabetes | 6 months
  The glycemic control will be measured by the change from baseline Glycosylated hemoglobin A1c (HbA1c) at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Zohar Landau, MD, Principal Investigator — Assuta Hospital Systems
Locations (1):
- AssutaHA, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wood JR, Miller KM, Maahs DM, Beck RW, DiMeglio LA, Libman IM, Quinn M, Tamborlane WV, Woerner SE; T1D Exchange Clinic Network. Most youth with type 1 diabetes in the T1D Exchange Clinic Registry do not meet American Diabetes Association or International Society for Pediatric and Adolescent Diabetes clinical guidelines. Diabetes Care. 2013 Jul;36(7):2035-7. doi: 10.2337/dc12-1959. Epub 2013 Jan 22. PMID 23340893
- [Result] Juvenile Diabetes Research Foundation Continuous Glucose Monitoring Study Group; Tamborlane WV, Beck RW, Bode BW, Buckingham B, Chase HP, Clemons R, Fiallo-Scharer R, Fox LA, Gilliam LK, Hirsch IB, Huang ES, Kollman C, Kowalski AJ, Laffel L, Lawrence JM, Lee J, Mauras N, O'Grady M, Ruedy KJ, Tansey M, Tsalikian E, Weinzimer S, Wilson DM, Wolpert H, Wysocki T, Xing D. Continuous glucose monitoring and intensive treatment of type 1 diabetes. N Engl J Med. 2008 Oct 2;359(14):1464-76. doi: 10.1056/NEJMoa0805017. Epub 2008 Sep 8. PMID 18779236
- [Result] Tonella P, Fluck CE, Mullis PE. Metabolic control of type 1 diabetic patients followed at the University Children's Hospital in Berne: have we reached the goal? Swiss Med Wkly. 2010 Jul 16;140:w13057. doi: 10.4414/smw.2010.13057. eCollection 2010. PMID 20648399
- [Result] Jean AM, Hassoun A, Hughes J, Pomeranz C, Fennoy I, McMahon DJ, Oberfield SE. Utility of early insulin response and proinsulin to assess insulin resistance. J Pediatr. 2009 Dec;155(6):893-9. doi: 10.1016/j.jpeds.2009.06.002. Epub 2009 Jul 29. PMID 19643436